CLINICAL TRIAL: NCT06364774
Title: Phase 1/2 Study Evaluating the Safety and Efficacy of Gene Therapy Employing Lentiviral Vector ALS20-transduced Hematopoietic Progenitor Cells in Subjects With Transfusion-dependent-thalassemia
Brief Title: ALS20-101 Lentiviral Gene Therapy for Beta Thalassemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-020309
Record Dates: First submitted 2024-03-26; First posted 2024-04-15 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Beta-Thalassemia
Keywords: Thalassemia; Beta Thalassemia; gene therapy; beta globin gene
MeSH Terms: conditions — beta-Thalassemia; Thalassemia

STUDY DESIGN:
Intervention Model Description: Single arm pilot, phase I/II study of 12 subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- beta thalassemia (Experimental): This arm will evaluate the safety and efficacy of infusing autologous hematopoietic stem and progenitor cells (HSPC) transduced with the novel lentiviral vector ALS20 that encodes the human βA-T87Q-globin gene, following myeloablative conditioning with busulfan.
  Interventions: Biological: ALS20

INTERVENTIONS:
Biological: ALS20 — novel lentiviral vector ALS20

SUMMARY:
The main goal of this study is to find out if the blood disorder called transfusion-dependent beta thalassemia can be safely treated by modifying blood stem cells. This is done by collecting blood stem cells from the subject, modifying those cells, adding a healthy beta globin gene, and then giving them back to the subject. It is hoped that these modified cells will decrease the need for blood transfusions. The gene modified blood stem cells are called CHOP-ALS20 ("study drug"). This experimental gene therapy has not been tried on human beings before and is not FDA approved.

DETAILED DESCRIPTION:
Beta thalassemia major is a hereditary blood disorder that requires lifelong regular transfusions and is associated with significant morbidity, early mortality, and decreased quality of life. Allogeneic hematopoietic stem cell transplantation is potentially curative but limited availability of suitable donors as well as risks of graft versus host disease limit its applicability. Gene addition of a functional beta globin gene may be an alternative treatment option.

The primary objective is to assess the safety of treatment with autologous hematopoietic stem cells transduced with a novel lentiviral vector (ALS20) in subjects 18 to <36 years old with transfusion dependent beta thalassemia.

The secondary objective is to evaluate the efficacy of treatment with autologous hematopoietic stem cells transduced with a novel lentiviral vector (ALS20) in subjects 18 to < 36 years old with transfusion dependent beta thalassemia.

Study Design: This is a single arm pilot, phase 1/2 study of up to 12 subjects ages 18 to <36 years who have transfusion-dependent beta thalassemia (genotypes β0β0, β+β0, β+β+, βEβ0, βEβ+, dominant β thalassemia). The study will evaluate the safety and efficacy of infusing autologous hematopoietic stem and progenitor cells (HSPC) transduced with the novel lentiviral vector ALS20 that encodes the human βA-T87Q-globin, following myeloablative conditioning with busulfan.

The main risks of this study involve risks of the genetic modification of the stem cells and the busulfan chemotherapy conditioning. Genetic modification of blood stem cells may increase the risk of blood cancer. The main risks of busulfan conditioning include prolonged low blood counts, liver injury, infertility, and cancer. There also is a risk of failure of the modified blood stem cells to grow.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to < 36 years at the time of consent
2. Diagnosis of transfusion dependent beta thalassemia (β0 β0, β+β0, β+β+, βEβ0, βEβ+,β0 or β+ /βA + alpha triplication(s)). Transfusion-dependent is defined as a history of receiving at least 120 mL/kg/year packed red blood cells or at least 8 transfusions per year in the past two years. The first 2 subjects enrolled must have a non- β0 β0 genotype.
3. Genetic confirmation of α and β thalassemia diagnosis (β0β0, β+β0, β+β+, βEβ0, βEβ+, β0 or β+ /βA + alpha triplication(s)) by a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory is required.
4. Clinically stable, Karnofsky score at least 70, and eligible to undergo Hematopoietic Stem Cell Transplantation (HSCT).
5. Female subjects of childbearing potential must agree to use acceptable method(s) of contraception from consent through at least 6 months after CHOP-ALS20 infusion
6. Male subjects of reproductive capacity must agree to use effective contraception from start of mobilization through at least 6 months after CHOP-ALS20 infusion
7. All potential treatment options including allogeneic HSCT (HLA-matched related, HLA-matched unrelated, and haploidentical) as well as FDA approved gene therapy options have been thoroughly discussed with the independent hematologist and/or transplant physician and subject agrees to proceed with this clinical trial.

Exclusion Criteria:

1. Prior receipt of HSCT or gene therapy
2. More than one alpha globin gene deletions/mutations.
3. Any prior or current malignancy (excluding adequately treated basal or squamous cell carcinoma of the skin)
4. Known cancer predisposition syndrome
5. Positive for HIV-1, HIV-2, Human T Cell Lymphotropic Virus-1,2 (HTLV-1, HTLV-2) or active hepatitis B or active hepatitis C infection
6. Clinically significant active bacterial, viral (including COVID-19 and influenza), fungal, or parasitic infection (temporary exclusion)
7. Clinically significant bleeding disorder
8. Evidence of cardiac dysfunction (left ventricular ejection fraction <50% or shortening fraction <27%) or clinically significant arrhythmia
9. Evidence of advanced liver disease (ALT >5x the upper limit of normal (ULN), prothrombin time >1.5 x ULN, direct bilirubin > 3x ULN) not attributable to iron chelation therapy, or evidence of bridging fibrosis on liver biopsy or fibrosis stage of F3 or higher by magnetic resonance elastography (MRE) if obtained as part of clinical care
10. Liver R2 or R2 MRI or liver biopsy with liver iron concentration 15 mg/g dw (temporary exclusion)
11. Diffusion capacity of the lungs for carbon monoxide (DLco) <50% of predicted (corrected for Hb)
12. Pulse oximetry in room air <92%
13. Evidence of renal dysfunction (creatinine >1.5x ULN or Glomerular Filtration Rate (GFR) <70 ml/min/1.73 m2 based on cystatin C/creatinine equation)
14. Cardiac T2 MRI < 10 ms
15. Platelet count <100,000/mcL or absolute neutrophil count <1000/mcL except if attributed to benign ethnic neutropenia
16. Unable to receive red cell transfusion (significant allo/auto immunization)
17. Uncontrolled systemic hypertension
18. Uncontrolled seizure disorder
19. Diagnosis of a significant psychiatric disorder that could seriously impede the ability to participate in the study as determined by the investigator
20. Immediate family member with a known or suspected Familial Cancer Syndrome
21. Contraindication to anesthesia
22. For female subjects, pregnancy or breastfeeding
23. Participation in another clinical trial of an investigational drug within 30 days or 5 drug half-lives, whichever is longer, of screening (temporary exclusion)
24. Any other condition that would render the subject ineligible for mobilization/apheresis and/or HSCT as determined by the investigator

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Neutrophil Engraftment | within 42 days after infusion
  time to neutrophil engraftment
Platelet Engraftment | through end of treatment, an average 1 year
  time to platelet engraftment
Overall Survival at 2 years | 2 years after treatment ends
  Survival status after treatment ends
Incidence of transplant related mortality | 1 year after infusion
  Incidence of transplant related mortality within 100 days and within 1 year after infusion
Incidence of Graft Versus Host Disease | through end of treatment, an average of 1 year
  any clinical evidence of graft versus host disease (GVHD)
Incidence of Vector-Derived Replication Competent Lentivirus | through end of treatment, an average of 1 year
  The detection of vector-derived replication competent lentivirus in any subject throughout the study until end of treatment.
Insertional Oncogenesis | through the end of the study, up to 24 months
  The number of subjects with insertional oncogenesis
Clonal Predominance | through the end of the study, up to 24 months
  The number of subjects with clonal predominance
maintain total hemoglobin level of 9.0 g/dL or higher | through the end of the study, up to 24 months
  The proportion of subjects able to discontinue regular red cell transfusions and maintain total hemoglobin level of 9.0 g/dL or higher (average over 1-year period) in the absence of red cell transfusion(transfusion independence). Success is defined as a minimum of 4 to 6 subjects achieving this endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Kwiatkowski, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No